CLINICAL TRIAL: NCT02879786
Title: Study of Hierarchy of Afferents in Postural Control of Children With Dyslexia
Acronym: EQUIDYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00139-32
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phonological dyslexia (Experimental): Children with phonological dyslexia
  Interventions: Other: Posturographic tests; Other: Questionnaire of motion sickness susceptibility
- Visuo-attentional dyslexia (Experimental): Children with visuo-attentional dyslexia
  Interventions: Other: Posturographic tests; Other: Questionnaire of motion sickness susceptibility
- Control (Other): Control children, age-matched
  Interventions: Other: Posturographic tests; Other: Questionnaire of motion sickness susceptibility

INTERVENTIONS:
Other: Posturographic tests
Other: Questionnaire of motion sickness susceptibility

SUMMARY:
The purpose is to determine the hierarchy of sensory afferents according to different forms of dyslexia in children.

The secondary purpose is to determine sensitive and sufficiently specific posturographic indexes for standard diagnosis of different types of dyslexia.

DETAILED DESCRIPTION:
This study evaluates the postural control and the importance of proprioception, evaluated by static and dynamic posturography, in dyslexic children compared to age-matched control group. Posturographic data and a questionnaire for motion sickness disorder are used as proprioceptive disorder index. This study aims to better characterize the dyslexic population with techniques targeting central integration of sensory proprioceptive afferents. The purpose of this study is not to search for a postural deficiency syndrome, but to study proprioception with posturography, with quantitative and normalized data of analyzed population. Moreover, these data could allow an objective evaluation of reeducation with quantifiable and reproducible parameters in order to judge its effectiveness. The demonstration of the existence of a relationship between proprioceptive disorders and dyslexia will imply a specific reeducation care of patients. A study using validated and standard indexes is necessary. The presence of postural disorders and a major susceptibility to motion sickness could contribute to distinguish different forms of dyslexia and thus be complementary to actual medical, orthophonic and neuropsychological criteria. In this evaluation, it is important to distinguish between visuo-attentional dyslexia from phonological dyslexia involving distinct anatomo-functional neuronal circuits.

ELIGIBILITY:
Inclusion Criteria:

All:

* Parents of child and child having given informed consent
* Affiliation to social security
* Preliminary medical examination

Dyslexia groups:

- Diagnosed and characterized dyslexia

Exclusion Criteria:

All:

* Medical pathology, especially neurological, ophthalmological, otorhinolaryngological or orthopedic, modifying postural control, detected with medical examination
* Insufficient compliance of child especially due to fatigue
* Contact allergy to cutaneous electrodes
* Current treatments: psychotropic drugs and all drugs diminishing awareness or causing dizziness or equilibrium disorders

Control group:

- Patient having a dyslexia or oral or written language disorder

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Score of evaluation of motion sickness susceptibility | day 0
Score of equilibrium evaluated with posturographic test | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PERRIN, Pr, Principal Investigator — INSERM U954 and Consultation ORL, Hôpital d'Enfants - CHU de Nancy
Locations (1):
- Centre de Référence pour les Troubles des Apprentissages - Hôpital d'Enfants - CHU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No